CLINICAL TRIAL: NCT01040624
Title: A Phase II Study of Proton-Based Radiation Therapy With Elective Pelvic Nodal Irradiation, Concomitant Docetaxel, and Adjuvant Androgen Deprivation for High-Risk Prostate Adenocarcinoma
Brief Title: Docetaxel, Androgen Deprivation and Proton Therapy for High Risk Prostate Cancer
Acronym: PR05
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 0703 - PR05; IRB201702459 (Other: UF IRB (New Number))
Record Dates: First submitted 2009-12-24; First posted 2009-12-29 (Estimated); Results first posted 2015-07-22 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer, Proton Radiation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-risk arm A (HR-A) (Experimental): < 15% risk of + lymph nodes (LN)
  Interventions: Radiation: < 15% risk of + LN
- HR-B (Experimental): > 15% risk of + LN
  Interventions: Radiation: > 15% risk of + LN

INTERVENTIONS:
Radiation: < 15% risk of + LN — Total of 54 Cobalt gray equivalent (CGE) over 30 treatments to prostate + seminal vesicles (SV), then proton boost total of 23.4-27 CGE over 13-15 treatments to prostate +/- SV. Low dose docetaxel every week during radiation therapy (RT) followed by androgen deprivation therapy for 6 months.
  Arms: High-risk arm A (HR-A)
Radiation: > 15% risk of + LN — Total of 45 Gy over 25 treatments to prostate + SV + LN, then proton boost total of 32.4-36 CGE over 18-20 treatments to prostate + SV. Low dose docetaxel every week during RT followed by androgen deprivation therapy for 6 months.
  Arms: HR-B

SUMMARY:
The purpose of this study is to see what effects, good and/or bad, proton based radiation combined with low dose chemotherapy and hormonal therapy, has on patients and their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the prostate.

Exclusion Criteria:

* Previous prostate cancer treatment such as chemotherapy and/or pelvic radiation.
* Active inflammatory bowel disease (diverticulitis, Crohn's disease or ulcerative colitis) affecting the rectum. (Non-active diverticulitis and Crohn's disease not affecting the rectum are allowed.)
* History of hip replacement.
* Prior intrapelvic surgery. This includes the following:
* Transrectal or rectal surgery other than polypectomy or hemorrhoid removal or banding
* Transabdominal pelvic surgery
* Bladder surgery
* Prior myocardial infarction (MI) or congestive heart failure (CHF).
* Taking Saw Palmetto or methotrexate and unable or unwilling to discontinue its use during radiation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-12; Primary Completion 2015-01 (Actual); Study Completion 2022-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy P Mendenhall, MD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

REFERENCES:
- [Background] American Joint Committee on Cancer. AJCC Cancer Staging Handbook, 6th ed. New York: Springer Verlag; 2002.
- [Background] Mendenhall NP, Li X, Morris CG, Keole S, Mendenhall WM, Nichols RC, Vargas C, Henderson RH, Early GI and GU toxicity in 3 prospective proton therapy trials for prostate cancer. Presented at the American Society of Therapeutic Radiation Oncologists. Chicago, 2009.
- [Background] Aizer AA, Yu JB, McKeon AM, Decker RH, Colberg JW, Peschel RE. Whole pelvic radiotherapy versus prostate only radiotherapy in the management of locally advanced or aggressive prostate adenocarcinoma. Int J Radiat Oncol Biol Phys. 2009 Dec 1;75(5):1344-9. doi: 10.1016/j.ijrobp.2008.12.082. Epub 2009 May 21. PMID 19464821
- [Background] Michalski JM, Bae K, Roach M, Markoe AM, Sandler HM, Ryu J, Parliament MB, Straube W, Valicenti RK, Cox JD. Long-term toxicity following 3D conformal radiation therapy for prostate cancer from the RTOG 9406 phase I/II dose escalation study. Int J Radiat Oncol Biol Phys. 2010 Jan 1;76(1):14-22. doi: 10.1016/j.ijrobp.2009.01.062. PMID 19577865
- [Background] Zelefsky MJ, Levin EJ, Hunt M, Yamada Y, Shippy AM, Jackson A, Amols HI. Incidence of late rectal and urinary toxicities after three-dimensional conformal radiotherapy and intensity-modulated radiotherapy for localized prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Mar 15;70(4):1124-9. doi: 10.1016/j.ijrobp.2007.11.044. PMID 18313526
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Schultz D, Blank K, Broderick GA, Tomaszewski JE, Renshaw AA, Kaplan I, Beard CJ, Wein A. Biochemical outcome after radical prostatectomy, external beam radiation therapy, or interstitial radiation therapy for clinically localized prostate cancer. JAMA. 1998 Sep 16;280(11):969-74. doi: 10.1001/jama.280.11.969. PMID 9749478
- [Background] Cox JD, Kian AK. Mosby Radiation Oncology: Rationale, Technique, Results, 8th ed.C.V. Mosby; 2002.
- [Background] Chism DB, Hanlon AL, Horwitz EM, Feigenberg SJ, Pollack A. A comparison of the single and double factor high-risk models for risk assignment of prostate cancer treated with 3D conformal radiotherapy. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):380-5. doi: 10.1016/j.ijrobp.2003.10.059. PMID 15145151
- [Background] Martinez AA, Demanes DJ, Galalae R, Vargas C, Bertermann H, Rodriguez R, Gustafson G, Altieri G, Gonzalez J. Lack of benefit from a short course of androgen deprivation for unfavorable prostate cancer patients treated with an accelerated hypofractionated regime. Int J Radiat Oncol Biol Phys. 2005 Aug 1;62(5):1322-31. doi: 10.1016/j.ijrobp.2004.12.053. PMID 16029788
- [Background] Roach M, Lu J, Pilepich MV, Asbell SO, Mohiuddin M, Terry R, Grignon D. Four prognostic groups predict long-term survival from prostate cancer following radiotherapy alone on Radiation Therapy Oncology Group clinical trials. Int J Radiat Oncol Biol Phys. 2000 Jun 1;47(3):609-15. doi: 10.1016/s0360-3016(00)00578-2. PMID 10837943
- [Background] Anaya-Saavedra G, Ramirez-Amador V, Irigoyen-Camacho ME, Garcia-Cuellar CM, Guido-Jimenez M, Mendez-Martinez R, Garcia-Carranca A. High association of human papillomavirus infection with oral cancer: a case-control study. Arch Med Res. 2008 Feb;39(2):189-97. doi: 10.1016/j.arcmed.2007.08.003. Epub 2007 Nov 8. PMID 18164962
- [Background] Partin AW, Mangold LA, Lamm DM, Walsh PC, Epstein JI, Pearson JD. Contemporary update of prostate cancer staging nomograms (Partin Tables) for the new millennium. Urology. 2001 Dec;58(6):843-8. doi: 10.1016/s0090-4295(01)01441-8. PMID 11744442
- [Background] Makarov DV, Trock BJ, Humphreys EB, Mangold LA, Walsh PC, Epstein JI, Partin AW. Updated nomogram to predict pathologic stage of prostate cancer given prostate-specific antigen level, clinical stage, and biopsy Gleason score (Partin tables) based on cases from 2000 to 2005. Urology. 2007 Jun;69(6):1095-101. doi: 10.1016/j.urology.2007.03.042. PMID 17572194
- [Background] Soloway MS, Pareek K, Sharifi R, Wajsman Z, McLeod D, Wood DP Jr, Puras-Baez A; Lupron Depot Neoadjuvant Prostate Cancer Study Group. Neoadjuvant androgen ablation before radical prostatectomy in cT2bNxMo prostate cancer: 5-year results. J Urol. 2002 Jan;167(1):112-6. PMID 11743286
- [Background] Hull GW, Rabbani F, Abbas F, Wheeler TM, Kattan MW, Scardino PT. Cancer control with radical prostatectomy alone in 1,000 consecutive patients. J Urol. 2002 Feb;167(2 Pt 1):528-34. doi: 10.1016/S0022-5347(01)69079-7. PMID 11792912
- [Background] Kestin LL, Martinez AA, Stromberg JS, Edmundson GK, Gustafson GS, Brabbins DS, Chen PY, Vicini FA. Matched-pair analysis of conformal high-dose-rate brachytherapy boost versus external-beam radiation therapy alone for locally advanced prostate cancer. J Clin Oncol. 2000 Aug;18(15):2869-80. doi: 10.1200/JCO.2000.18.15.2869. PMID 10920135
- [Background] Demanes DJ, Rodriguez RR, Schour L, Brandt D, Altieri G. High-dose-rate intensity-modulated brachytherapy with external beam radiotherapy for prostate cancer: California endocurietherapy's 10-year results. Int J Radiat Oncol Biol Phys. 2005 Apr 1;61(5):1306-16. doi: 10.1016/j.ijrobp.2004.08.014. PMID 15817332
- [Background] Pickles T, Keyes M, Morris WJ. Brachytherapy or conformal external radiotherapy for prostate cancer: a single-institution matched-pair analysis. Int J Radiat Oncol Biol Phys. 2010 Jan 1;76(1):43-9. doi: 10.1016/j.ijrobp.2009.01.081. PMID 19570619
- [Background] Roach M 3rd, DeSilvio M, Lawton C, Uhl V, Machtay M, Seider MJ, Rotman M, Jones C, Asbell SO, Valicenti RK, Han S, Thomas CR Jr, Shipley WS; Radiation Therapy Oncology Group 9413. Phase III trial comparing whole-pelvic versus prostate-only radiotherapy and neoadjuvant versus adjuvant combined androgen suppression: Radiation Therapy Oncology Group 9413. J Clin Oncol. 2003 May 15;21(10):1904-11. doi: 10.1200/JCO.2003.05.004. PMID 12743142
- [Background] Lawton CA, DeSilvio M, Roach M 3rd, Uhl V, Kirsch R, Seider M, Rotman M, Jones C, Asbell S, Valicenti R, Hahn S, Thomas CR Jr. An update of the phase III trial comparing whole pelvic to prostate only radiotherapy and neoadjuvant to adjuvant total androgen suppression: updated analysis of RTOG 94-13, with emphasis on unexpected hormone/radiation interactions. Int J Radiat Oncol Biol Phys. 2007 Nov 1;69(3):646-55. doi: 10.1016/j.ijrobp.2007.04.003. Epub 2007 May 24. PMID 17531401
- [Background] Pommier P, Chabaud S, Lagrange JL, Richaud P, Lesaunier F, Le Prise E, Wagner JP, Hay MH, Beckendorf V, Suchaud JP, Pabot du Chatelard PM, Bernier V, Voirin N, Perol D, Carrie C. Is there a role for pelvic irradiation in localized prostate adenocarcinoma? Preliminary results of GETUG-01. J Clin Oncol. 2007 Dec 1;25(34):5366-73. doi: 10.1200/JCO.2006.10.5171. PMID 18048817
- [Background] Zietman AL, DeSilvio ML, Slater JD, Rossi CJ Jr, Miller DW, Adams JA, Shipley WU. Comparison of conventional-dose vs high-dose conformal radiation therapy in clinically localized adenocarcinoma of the prostate: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1233-9. doi: 10.1001/jama.294.10.1233. PMID 16160131
- [Background] Sathya JR, Davis IR, Julian JA, Guo Q, Daya D, Dayes IS, Lukka HR, Levine M. Randomized trial comparing iridium implant plus external-beam radiation therapy with external-beam radiation therapy alone in node-negative locally advanced cancer of the prostate. J Clin Oncol. 2005 Feb 20;23(6):1192-9. doi: 10.1200/JCO.2005.06.154. PMID 15718316
- [Background] Dearnaley DP, Hall E, Lawrence D, Huddart RA, Eeles R, Nutting CM, Gadd J, Warrington A, Bidmead M, Horwich A. Phase III pilot study of dose escalation using conformal radiotherapy in prostate cancer: PSA control and side effects. Br J Cancer. 2005 Feb 14;92(3):488-98. doi: 10.1038/sj.bjc.6602301. PMID 15685244
- [Background] Shipley WU, Verhey LJ, Munzenrider JE, Suit HD, Urie MM, McManus PL, Young RH, Shipley JW, Zietman AL, Biggs PJ, et al. Advanced prostate cancer: the results of a randomized comparative trial of high dose irradiation boosting with conformal protons compared with conventional dose irradiation using photons alone. Int J Radiat Oncol Biol Phys. 1995 Apr 30;32(1):3-12. doi: 10.1016/0360-3016(95)00063-5. PMID 7721636
- [Background] Kuban DA, Tucker SL, Dong L, Starkschall G, Huang EH, Cheung MR, Lee AK, Pollack A. Long-term results of the M. D. Anderson randomized dose-escalation trial for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):67-74. doi: 10.1016/j.ijrobp.2007.06.054. Epub 2007 Aug 31. PMID 17765406
- [Background] Pollack A, Hanlon AL, Horwitz EM, Feigenberg SJ, Uzzo RG, Hanks GE. Prostate cancer radiotherapy dose response: an update of the fox chase experience. J Urol. 2004 Mar;171(3):1132-6. doi: 10.1097/01.ju.0000111844.95024.74. PMID 14767286
- [Background] Fuks Z, Leibel SA, Wallner KE, Begg CB, Fair WR, Anderson LL, Hilaris BS, Whitmore WF. The effect of local control on metastatic dissemination in carcinoma of the prostate: long-term results in patients treated with 125I implantation. Int J Radiat Oncol Biol Phys. 1991 Aug;21(3):537-47. doi: 10.1016/0360-3016(91)90668-t. PMID 1869452
- [Background] Vargas C, Martinez A, Boike TP, Edmundson G, Gustafson G, Krauss D. Long Term Survival Benefit of a Prospective Dose Escalation Trial Using High Dose Rate (HDR) Brachytherapy Boost. [Abstr.] Int J Radiat Oncol Biol Phys 2005;63:S37-S38.
- [Background] Vargas C, Fryer A, Mahajan C, Indelicato D, Horne D, Chellini A, McKenzie C, Lawlor P, Henderson R, Li Z, Lin L, Olivier K, Keole S. Dose-volume comparison of proton therapy and intensity-modulated radiotherapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Mar 1;70(3):744-51. doi: 10.1016/j.ijrobp.2007.07.2335. Epub 2007 Sep 27. PMID 17904306
- [Background] Zietman AL. Correction: Inaccurate analysis and results in a study of radiation therapy in adenocarcinoma of the prostate. JAMA. 2008 Feb 27;299(8):898-9. doi: 10.1001/jama.299.8.898-c. No abstract available. PMID 18314431
- [Background] Karakiewicz PI, Bhojani N, Capitanio U, Reuther AM, Suardi N, Jeldres C, Pharand D, Peloquin F, Perrotte P, Shariat SF, Klein EA. External validation of the updated Partin tables in a cohort of North American men. J Urol. 2008 Sep;180(3):898-902; discussion 902-3. doi: 10.1016/j.juro.2008.05.044. Epub 2008 Jul 17. PMID 18635222
- [Background] Bastide C, Brenot-Rossi I, Garcia S, Rossi D. Radioisotope guided sentinel lymph node dissection in patients with localized prostate cancer: results of the first 100 cases. Eur J Surg Oncol. 2009 Jul;35(7):751-6. doi: 10.1016/j.ejso.2008.04.007. Epub 2008 Jun 6. PMID 18538526
- [Background] Winter A, Wawroschek F. Lymphadenectomy in prostate cancer. Radio-guided lymph node mapping: an adequate staging method. Front Radiat Ther Oncol. 2008;41:58-67. doi: 10.1159/000139879. PMID 18544986
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] Petrylak DP, Tangen CM, Hussain MH, Lara PN Jr, Jones JA, Taplin ME, Burch PA, Berry D, Moinpour C, Kohli M, Benson MC, Small EJ, Raghavan D, Crawford ED. Docetaxel and estramustine compared with mitoxantrone and prednisone for advanced refractory prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1513-20. doi: 10.1056/NEJMoa041318. PMID 15470214
- [Background] Chi KN, Chin JL, Winquist E, Klotz L, Saad F, Gleave ME. Multicenter phase II study of combined neoadjuvant docetaxel and hormone therapy before radical prostatectomy for patients with high risk localized prostate cancer. J Urol. 2008 Aug;180(2):565-70; discussion 570. doi: 10.1016/j.juro.2008.04.012. Epub 2008 Jun 12. PMID 18554663
- [Background] Kumar P, Perrotti M, Weiss R, Todd M, Goodin S, Cummings K, DiPaola RS. Phase I trial of weekly docetaxel with concurrent three-dimensional conformal radiation therapy in the treatment of unfavorable localized adenocarcinoma of the prostate. J Clin Oncol. 2004 May 15;22(10):1909-15. doi: 10.1200/JCO.2004.02.001. PMID 15143084
- [Background] Bolla M, Collette L, Blank L, Warde P, Dubois JB, Mirimanoff RO, Storme G, Bernier J, Kuten A, Sternberg C, Mattelaer J, Lopez Torecilla J, Pfeffer JR, Lino Cutajar C, Zurlo A, Pierart M. Long-term results with immediate androgen suppression and external irradiation in patients with locally advanced prostate cancer (an EORTC study): a phase III randomised trial. Lancet. 2002 Jul 13;360(9327):103-6. doi: 10.1016/s0140-6736(02)09408-4. PMID 12126818
- [Background] Crook J, Ludgate C, Malone S, Lim J, Perry G, Eapen L, Bowen J, Robertson S, Lockwood G. Report of a multicenter Canadian phase III randomized trial of 3 months vs. 8 months neoadjuvant androgen deprivation before standard-dose radiotherapy for clinically localized prostate cancer. Int J Radiat Oncol Biol Phys. 2004 Sep 1;60(1):15-23. doi: 10.1016/j.ijrobp.2004.02.022. PMID 15337535
- [Background] D'Amico AV, Manola J, Loffredo M, Renshaw AA, DellaCroce A, Kantoff PW. 6-month androgen suppression plus radiation therapy vs radiation therapy alone for patients with clinically localized prostate cancer: a randomized controlled trial. JAMA. 2004 Aug 18;292(7):821-7. doi: 10.1001/jama.292.7.821. PMID 15315996
- [Background] Hanks GE, Pajak TF, Porter A, Grignon D, Brereton H, Venkatesan V, Horwitz EM, Lawton C, Rosenthal SA, Sandler HM, Shipley WU; Radiation Therapy Oncology Group. Phase III trial of long-term adjuvant androgen deprivation after neoadjuvant hormonal cytoreduction and radiotherapy in locally advanced carcinoma of the prostate: the Radiation Therapy Oncology Group Protocol 92-02. J Clin Oncol. 2003 Nov 1;21(21):3972-8. doi: 10.1200/JCO.2003.11.023. PMID 14581419
- [Background] Pilepich MV, Winter K, John MJ, Mesic JB, Sause W, Rubin P, Lawton C, Machtay M, Grignon D. Phase III radiation therapy oncology group (RTOG) trial 86-10 of androgen deprivation adjuvant to definitive radiotherapy in locally advanced carcinoma of the prostate. Int J Radiat Oncol Biol Phys. 2001 Aug 1;50(5):1243-52. doi: 10.1016/s0360-3016(01)01579-6. PMID 11483335
- [Background] Pilepich MV, Winter K, Lawton CA, Krisch RE, Wolkov HB, Movsas B, Hug EB, Asbell SO, Grignon D. Androgen suppression adjuvant to definitive radiotherapy in prostate carcinoma--long-term results of phase III RTOG 85-31. Int J Radiat Oncol Biol Phys. 2005 Apr 1;61(5):1285-90. doi: 10.1016/j.ijrobp.2004.08.047. PMID 15817329
- [Background] D'Amico AV, Loffredo M, Renshaw AA, Loffredo B, Chen MH. Six-month androgen suppression plus radiation therapy compared with radiation therapy alone for men with prostate cancer and a rapidly increasing pretreatment prostate-specific antigen level. J Clin Oncol. 2006 Sep 1;24(25):4190-5. doi: 10.1200/JCO.2006.06.8239. PMID 16943536
- [Background] Denham JW, Steigler A, Wilcox C, Lamb DS, Joseph D, Atkinson C, Matthews J, Tai KH, Spry NA, Christie D, Gleeson PS, Greer PB, D'Este C; Trans-Tasman Radiation Oncology Group 96.01 Trialists. Time to biochemical failure and prostate-specific antigen doubling time as surrogates for prostate cancer-specific mortality: evidence from the TROG 96.01 randomised controlled trial. Lancet Oncol. 2008 Nov;9(11):1058-68. doi: 10.1016/S1470-2045(08)70236-5. Epub 2008 Oct 15. PMID 18929505
- [Background] Bolla M, de Reijke TM, Van Tienhoven G, Van den Bergh AC, Oddens J, Poortmans PM, Gez E, Kil P, Akdas A, Soete G, Kariakine O, van der Steen-Banasik EM, Musat E, Pierart M, Mauer ME, Collette L; EORTC Radiation Oncology Group and Genito-Urinary Tract Cancer Group. Duration of androgen suppression in the treatment of prostate cancer. N Engl J Med. 2009 Jun 11;360(24):2516-27. doi: 10.1056/NEJMoa0810095. PMID 19516032
- [Background] Ghilezan MJ, Jaffray DA, Siewerdsen JH, Van Herk M, Shetty A, Sharpe MB, Zafar Jafri S, Vicini FA, Matter RC, Brabbins DS, Martinez AA. Prostate gland motion assessed with cine-magnetic resonance imaging (cine-MRI). Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):406-17. doi: 10.1016/j.ijrobp.2003.10.017. PMID 15890582
- [Background] Padhani AR, Khoo VS, Suckling J, Husband JE, Leach MO, Dearnaley DP. Evaluating the effect of rectal distension and rectal movement on prostate gland position using cine MRI. Int J Radiat Oncol Biol Phys. 1999 Jun 1;44(3):525-33. doi: 10.1016/s0360-3016(99)00040-1. PMID 10348281
- [Background] Litzenberg D, Dawson LA, Sandler H, Sanda MG, McShan DL, Ten Haken RK, Lam KL, Brock KK, Balter JM. Daily prostate targeting using implanted radiopaque markers. Int J Radiat Oncol Biol Phys. 2002 Mar 1;52(3):699-703. doi: 10.1016/s0360-3016(01)02654-2. PMID 11849792
- [Background] Litzenberg DW, Balter JM, Hadley SW, Sandler HM, Willoughby TR, Kupelian PA, Levine L. Influence of intrafraction motion on margins for prostate radiotherapy. Int J Radiat Oncol Biol Phys. 2006 Jun 1;65(2):548-53. doi: 10.1016/j.ijrobp.2005.12.033. Epub 2006 Mar 20. PMID 16545919
- [Background] Vargas C, Yan D, Kestin LL, Krauss D, Lockman DM, Brabbins DS, Martinez AA. Phase II dose escalation study of image-guided adaptive radiotherapy for prostate cancer: use of dose-volume constraints to achieve rectal isotoxicity. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):141-9. doi: 10.1016/j.ijrobp.2004.12.017. PMID 16111582

RESULTS

PARTICIPANT FLOW:
Groups:
- HR-A: < 15% risk of + lymph nodes (LN)
  < 15% risk of + LN: Total of 54 Cobalt gray equivalent (CGE) over 30 treatments to prostate + seminal vesicles (SV), then proton boost total of 23.4-27 CGE over 13-15 treatments to prostate +/- SV. Low dose docetaxel every week during radiation therapy (RT) followed by androgen deprivation therapy for 6 months.
Period: Overall Study
Arm/Group | HR-A | HR-B
Started | 58 | 19
Completed | 58 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HR-A: < 15% risk of + LN
  < 15% risk of + LN: Total of 54 CGE over 30 treatments to prostate + SV, then proton boost total of 23.4-27 CGE over 13-15 treatments to prostate +/- SV. Low dose docetaxel every week during RT followed by androgen deprivation therapy for 6 months.
- Total: Total of all reporting groups
Arm/Group | HR-A | HR-B | Total
Number analyzed (Participants) | 58 | 19 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 4 | 20
  >=65 years | 42 | 15 | 57
Age, Continuous [Median (Full Range); unit: years] | 68 [52 to 80] | 69 [51 to 79] | 68 [51 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 58 | 19 | 77
Region of Enrollment [Number; unit: participants]
  United States | 58 | 19 | 77

OUTCOME MEASURES:

1. Primary Outcome: Acute Grade 3 or Higher Treatment-related Toxicity Rate.
Description: Number of participants that experienced acute grade 3 or higher, treatment-related toxicity based on CTCAE version 3.0 criteria.
Time Frame: 6 months after the completion of radiation therapy
Measure: Number; unit: participants
Arm/Group | HR-A | HR-B
Number analyzed (Participants) | 58 | 19
participants | 1 | 3
Statistical Analysis 1: Comparison: HR-A vs HR-B; Test type: Superiority or Other; p < 0.0001, Chi-squared; One-sided binomial test of univariate probability distributions

2. Secondary Outcome: Collect and Analyze Quality of Life, Treatment-related Late Morbidity, Disease Control, and Survival Outcome Parameters.
Time Frame: After radiation: every 6 months for 3 years, then annually for 20 years
Reporting Status: Not Posted

3. Secondary Outcome: Collect and Analyze Treatment, Biologic and Diagnostic Information That May Impact Quality of Life, Disease Control, Morbidity and/or Survival Outcomes.
Time Frame: After radiation: every 6 months for 3 years, then annually for 20 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | HR-A | HR-B
Serious Adverse Events (participants affected / at risk) | 1/58 | 3/19
Other Adverse Events (participants affected / at risk) | 13/58 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HR-A (N=58) | HR-B (N=19)
Diarrhea - acute (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation - acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal cramping - acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain - acute (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HR-A (N=58) | HR-B (N=19)
Pain - acute (General disorders) | 6 (6) | 2 (2)
Constipation - acute (Gastrointestinal disorders) | 5 (5) | 2 (2)
Diarrhea - acute (Gastrointestinal disorders) | 4 (4) | 7 (7)
Dysuria - acute (Renal and urinary disorders) | 3 (3) | 0 (0)
Abdominal cramping acute (Gastrointestinal disorders) | 1 (1) | 2 (2)
Obstruction - acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Proctitis - acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal bleeding - late (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal cramping - late (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation - late (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No